CLINICAL TRIAL: NCT06197269
Title: Efficacy And Safety Of Short Course Antibiotic Therapy (72hrs) As Compared To Standard Duration (5-7 Days) Of Therapy In Preterm Neonates With Culture Negative Early Onset Sepsis: A Randomized Controlled Trial
Brief Title: Efficacy And Safety Of Short Course Antibiotic Therapy In Preterm Neonates With Early Onset Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, Sushma Nangia, M.D., Director Professor & Head, Department of Neonatology, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LHMC/IEC/2019/41
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Early-Onset Neonatal Sepsis; Antibiotic Stewardship
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short duration antibiotic (Experimental): antibiotic therapy will be stopped at the time of randomization i.e. 72 hrs after starting treatment
  Interventions: Other: Short duration antibiotics
- Standard duration antibiotic (Active Comparator): Antibiotics will be continued for 5-7 days more, 72 hrs after starting treatment.
  Interventions: Other: Standard duration antibiotics

INTERVENTIONS:
Other: Short duration antibiotics — antibiotic therapy will be stopped at the time of randomization i.e. 72 hrs after starting treatment
  Arms: Short duration antibiotic
Other: Standard duration antibiotics — Antibiotics will be continued for 5-7 days more, 72 hrs after starting treatment.
  Arms: Standard duration antibiotic

SUMMARY:
Objective of the study is to compare the efficacy and safety of 'Short duration antibiotic' (72hrs) and 'Standard duration antibiotic'(5 - 7days) in preterm neonates ( >28weeks and >1000grams ) with culture negative early onset sepsis.

DETAILED DESCRIPTION:
Enrolled participants will be randomly allocated to one of two study groups: 1) Short duration antibiotic' (72hrs), 2) Standard duration antibiotic'(5 - 7days)

Short duration antibiotic group: Antibiotic therapy stopped at the time of randomization i.e. 72 hours after starting antibiotics

Standard duration antibiotic group: antibiotics therapy continued for 5-7 days further after 72 hrs of starting antibiotics.

ELIGIBILITY:
Inclusion Criteria (All must be present)

* All Preterm neonates (Gestational age >28weeks and >1000grams)
* age less than 72hours of life
* Started on antibiotic therapy based on presence of symptoms attributable to sepsis and /or positive sepsis screen but sterile blood culture
* Symptoms resolved at time of randomization

Exclusion Criteria:

* Antibiotics started based on risk factors
* Infants with major congenital anomalies or syndromes.
* Presence of site specific infections including meningitis, pneumonia
* Neonates suspected to have inborn errors of metabolism
* Neonates with Severe birth asphyxia, (Apgar score at 5min <4 and cord Ph< 7.0,base excess <-16)
* Neonates underwent major surgery in 1st week of life
* Deemed by Doctor in charge to be sick enough to be continued on antibiotics

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-04-14 (Actual)

PRIMARY OUTCOMES:
Incidence of 'Treatment Failure' | 15 days of stopping antibiotics
  New onset appearance of clinical signs and symptoms requiring initiation of antibiotics

SECONDARY OUTCOMES:
Mortality | Till 1 month of life
  Death due to any reason
Need for additional courses of antibiotic therapy | Till 1 month of life
  Additional courses during the study time frame
Length of hospital stay | From date of birth until date of death or discharge whichever come assessed till 1 month of life
  Duration of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Lady Hardinge Medical college, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No